CLINICAL TRIAL: NCT04937725
Title: Reading Problems Associated With Central Nervous System Pathologies
Brief Title: Reading Problems Associated With Central Nervous System (CNS) Pathologies.
Status: Completed | Type: Observational
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other); Hospital del Rio Hortega (Other)
Responsible Party: Sponsor
Other Study IDs: PI21-2247 TFM
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Injury Brain; Eye Abnormalities; Multiple Sclerosis; Parkinson Disease; Ataxia, Cerebellar
Keywords: eye tracking
MeSH Terms: conditions — Brain Injuries; Eye Abnormalities; Multiple Sclerosis; Parkinson Disease; Cerebellar Ataxia | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Patients without neurological pathologies: Patients with no history of neurological diseases
  Interventions: Diagnostic Test: eye tracking
- Patients with neurological pathologies
  Interventions: Diagnostic Test: eye tracking

INTERVENTIONS:
Diagnostic Test: eye tracking — Eye tracker will be used to evaluate study parameters

SUMMARY:
This project aims to analyse eye movements, their alterations and influence in reading performance in patients with acquired CNS diseases and compare them with people of the same age, without neurological or ocular pathology and with normal reading speed and pattern.

The exploration is focused on the oculomotor system in patients with CNS diseases, even without involvement of the primary visual pathway, and reveals more involvement than the one obtained by a simple ophthalmological examination.

DETAILED DESCRIPTION:
The following protocol will be applied:

Neuropsychological function Clock Test- Clock Drawing, whose score corresponds to a scale of 1 to 6, from perfect organization to severe disorder respectively, with a cognitive deficit being a result greater than 3. This test is used to detect signs of heminegligence in addition to the Line Bisection Test. It will consider the displacement of the central mark to the right side as a positive sign.

Mini-Cognitive Exam, whose cut-off score corresponds to 23 out of the 30 total, equal to or less than this figure, would indicate the presence of a cognitive deficit.

Far and near Best corrected visual acuity Primary gaze position Cover test (far and near) Extrinsic ocular motility Nystagmus presence Intrinsic ocular motility Biomicroscopy of the anterior pole Computerized visual field 30-2 Intraocular pressure Ocular fundus examination Records with Tobii Pro Nano Hardware Package eye-tracking system and Tobii Pro Lab - Full Edition software.

Reading performance assessment: International Reading Speed Texts (IReST) Attentional questionnaire based on the IReST, two simple answer questions (one word) will be formulated for each text, at the end of the reading to check the reading comprehension of the patient Evaluation of the speed and quality of horizontal and vertical reading: Test DEM (Developmental Eye Movement).

Eye-tracking test: with an animation of a moving circle.

ELIGIBILITY:
Inclusion Criteria:

* Patients and normal volunteers with ages between 18 and 80 years old.
* Clinical radiological neurological stability in acute CNS diseases (≥ 3 months after ACD).
* Best distant binocular visual acuity, equal or greater than 0.5 (Decimal Scale). Best close binocular visual acuity, equal or greater than 20/40.Glasses or soft contact lenses users.

Exclusion Criteria:

* Presence of visual heminegligence evaluated with clock drawing test and line bisection test.
* Presence of visual agnosia: Poppelreuter-Ghent © test.
* Presence of cognitive deficit: mini mental state examination (MMSE), with sufficient residual hearing capacity.
* Medical history, or presence after ophthalmic examination of: maculopathy, advanced cataracts, ophthalmological diseases affecting central visual acuity or macular fixation.
* Healthy control subjects should have normal monocular perimetry using standard Swedish interactive threshold algorithm (SITA) Central 30-2 Humphrey® Perimeter Test .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal population (no pathology) and people with neurological pathologies such as multiple sclerosis, Parkinson, tumours, or stroke, cerebellum ataxia and other miscellaneous neurological disorders.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Reading performance | 24 Hours
  International Reading Speed Texts (IReST)

SECONDARY OUTCOMES:
Reading performance | 24 Hours
  DEM (Developmental Eye Movement).ocular (DEM)

OTHER OUTCOMES:
Eye tracking | 24 Hours
  Eye-tracking test

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA - Universidad de Valladolid, Valladolid, Spain